CLINICAL TRIAL: NCT03741270
Title: Safety of Rabivax-S in Individuals Receiving Pre-exposure Prophylaxis (PrEP)
Brief Title: Safety of Rabivax-S for Pre-exposure Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ross University School of Veterinary Medicine (Other)
Collaborators: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Darryn Knobel, Professor of Epidemiology and Population Health, Ross University School of Veterinary Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-13-EX
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Rabies Vaccine Adverse Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine (Experimental)
  Interventions: Biological: Rabivax-S

INTERVENTIONS:
Biological: Rabivax-S — Rabivax-S is a lyophilized vaccine manufactured by Serum Institute of India Pvt. Ltd. containing inactivated purified rabies antigen (Pitman Moore, PM3218 as virus strain) produced using Vero ATCC CCL 81 cells. The diluent (sterile water for injection) is provided in a separate 1 mL ampoule. After reconstitution, a single dose of 1 mL contains an inactivated, purified rabies antigen (not less than 2.5 IU), glycine (40 mg), sucrose (40 mg) and human serum albumin (25% 10 mg). The intervention is administered by intramuscular injection of 1 mL reconstituted vaccine in the deltoid area of the upper arm, on days 0, 7 and 21 (or 28).

SUMMARY:
People who are at frequent or continuous risk of exposure to rabies virus should be vaccinated against the disease (pre-exposure prophylaxis). This includes people who work with rabies virus in research or diagnostic laboratories or vaccine production facilities, veterinarians, staff, animal-control and wildlife workers in areas where rabies is endemic. Veterinary students in clinical placements and externships are included in this category. Currently, DVM students at Ross University School of Veterinary Medicine (RUSVM) are vaccinated against rabies in their 7th semester (final pre-clinical semester). Vaccinations are done by RUSVM Health Services using Rabivax-S, produced by the Serum Institute of India (study co-sponsors). Previously-unvaccinated students receive three injections of vaccine, on day 0, 7 and 21-28. The aim of the study is to generate additional data on safety and tolerability of Rabivax-S administered as pre-exposure prophylaxis to this population.

ELIGIBILITY:
Inclusion Criteria:

A DVM student registered at RUSVM will be eligible for inclusion in the study if the student is:

1. in the 7th semester of the DVM program, or
2. is in the 5th or 6th semester of the DVM program and is planning to undertake a veterinary externship in the following semester break that would require pre-exposure prophylaxis to rabies.

Exclusion Criteria:

A DVM student who meets the inclusion criteria will be excluded from the study if the student:

1. has previously received a dose of rabies vaccine, or
2. has any condition for which rabies vaccination is contra-indicated, or
3. does not provide informed consent for participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with at least one solicited adverse event (AE) within 4 days after any dose | Through 4 days after each dose
  Based on the package insert for Rabivax-S, the following adverse events will be solicited:
  * Local reactions (limited to the site of the injection): pain, erythema, oedema, pruritus and induration.
  * Systemic reactions: fever, shivering, malaise, asthenia, faintness, dizziness, headache, myalgia, arthralgia, nausea and abdominal pain.
  * Hypersensitivity or allergic reactions: anaphylaxis, urticaria, rash and erythema multiforme.

SECONDARY OUTCOMES:
Number of unsolicited adverse events during 28 days after the first dose | Through 28 days after the first dose given (day 0)
  Definitions of AEs and SAEs are taken from the OHRP's Guidance on Reviewing and Reporting Unanticipated Problems Involving Risks to Subjects or Others and Adverse Events.
  AE means any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research.
  A SAE is any AE temporally associated with the subject's participation in research that meets any of the following criteria:
  1. results in death;
  2. is life-threatening;
  3. requires inpatient hospitalization;
  4. results in a persistent or significant disability/incapacity;
  5. results in a congenital anomaly/birth defect; or
  6. any other AE that, based upon appropriate medical judgment, may jeopardize the subject's health and may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of serious adverse events during 28 days after the first dose | Through 28 days after the first dose given (day 0)
Number of participants with at least one solicited adverse event (AE) within 4 days after first dose | Through 4 days after first dose (days 0-3)
Number of participants with at least one solicited adverse event (AE) within 4 days after second dose | Through 4 days after second dose (days 7-10)
Number of participants with at least one solicited adverse event (AE) within 4 days after third dose | Through 4 days after second dose (days 21-24 or days 28-31)

CONTACTS AND LOCATIONS:
Overall Officials: Darryn L Knobel, BVSc, PhD, Principal Investigator — Ross University School of Veterinary Medicine
Locations (1):
- Ross University School of Veterinary Medicine, Basseterre, Saint Kitts and Nevis

IPD SHARING:
Plan to Share IPD: Yes